CLINICAL TRIAL: NCT06784531
Title: The Influence of Race and MitoQ Supplementation on Skin Perfusion in the Cold
Brief Title: The Influence of Race and MitoQ Supplementation on Skin Blood Flow in the Cold
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 23-16H; MO230093 (Other Grant/Funding Number: U.S. Army Medical Research and Development Command)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Cold Exposure
Keywords: Skin blood flow; Skin temperature; Oxidative stress; Vasoconstriction; Cold stress; Racial disparities; Reactive oxygen species; Mitochondrial antioxidant; Mitoquinone; Mitoquinol; Manual dexterity; Peripheral cold injury
MeSH Terms: interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo - Cold Water Hand Immersion (Placebo Comparator): Four placebo (microcrystalline cellulose) capsules are taken ~1 hour before a 30-minute hand immersion in 54°F water.
  Interventions: Dietary Supplement: Placebo; Other: Cold Water Hand Immersion
- Placebo - Cold Air Exposure (Placebo Comparator): Four placebo (microcrystalline cellulose) capsules are taken ~1 hour before a 90-minute cold exposure in 41°F air.
  Interventions: Dietary Supplement: Placebo; Other: Cold Air Exposure
- MitoQ - Cold Water Hand Immersion (Experimental): Four 20 mg MitoQ capsules (80 mg total) are taken ~1 hour before a 30-minute hand immersion in 54°F water.
  Interventions: Dietary Supplement: Mitoquinone mesylate (MitoQ); Other: Cold Water Hand Immersion
- MitoQ - Cold Air Exposure (Experimental): Four 20 mg MitoQ capsules (80 mg total) are taken ~1 hour before a 90-minute cold exposure in 41°F air.
  Interventions: Dietary Supplement: Mitoquinone mesylate (MitoQ); Other: Cold Air Exposure

INTERVENTIONS:
Dietary Supplement: Mitoquinone mesylate (MitoQ) — Four 20 mg MitoQ capsules (80 mg total) are ingested orally.
  Arms: MitoQ - Cold Air Exposure; MitoQ - Cold Water Hand Immersion
Dietary Supplement: Placebo — Four placebo (microcrystalline cellulose) capsules are ingested orally.
  Arms: Placebo - Cold Air Exposure; Placebo - Cold Water Hand Immersion
Other: Cold Water Hand Immersion — Volunteers place one hand in cold (54°F) water for 30 minutes.
  Arms: MitoQ - Cold Water Hand Immersion; Placebo - Cold Water Hand Immersion
Other: Cold Air Exposure — Volunteers sit in cold (41°F) air for 90 minutes.
  Arms: MitoQ - Cold Air Exposure; Placebo - Cold Air Exposure

SUMMARY:
Individuals who operate in cold weather are at risk of developing cold injuries, for example, frostbite. They also often experience a loss of hand function and joint mobility due to a decrease in skin temperature and blood flow.

In addition, the risk of getting a cold injury is higher in the Black population compared to other racial and ethnic groups. Increases in oxidant compounds can cause the blood vessels in the skin to narrow and decrease skin temperature in the cold. However, it is unknown whether the higher risk of cold injury in Black individuals is because of a greater amount of oxidant compounds in the blood vessels. The purpose of this research is to see if an antioxidant supplement called MitoQ can help to improve skin temperature and blood flow in the cold and if the improvement is greater in Black individuals.

DETAILED DESCRIPTION:
In a randomized, double-blinded, crossover design, healthy volunteers (18-40 yrs) will undergo a set of cold exposures following acute ingestion of a high-dose MitoQ supplement and placebo. The cold exposures will consist of a hand immersion in 54°F water and a 90-min exposure to 41°F air during which skin blood flow and temperatures will be measured. The hypothesis is that the declines in skin blood flow and temperature will be greater during cold exposure in Black individuals and that MitoQ supplementation will improve skin blood flow and temperature to a greater extent in Black individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-40
* In good health as determined by OMSO (Office of Medical Support and Oversight)
* Willing to refrain from exercise and caffeinated or alcoholic beverages for 12 hours before each testing session
* Willing to refrain from antioxidant-rich foods, such as blueberries, pecans, and dark chocolate, 48 h before each testing session
* Eumenorrheic females (menstrual cycle length between 24-35 days) or females taking oral contraceptives, or utilizing implantable contraception (e.g., intrauterine device)
* Have supervisor approval if active-duty military or a federal employee at NSSC

Exclusion Criteria:

* History of cold injuries of any severity (e.g., frostbite, trench foot, chilblains)
* Raynaud's syndrome
* Cold-induced asthma/bronchospasm
* Previous hand/finger injuries that impair dexterity and hand function
* Metal hardware (plates/screws) in the forearms and hands
* Smoke, vape, or use smokeless tobacco or other nicotine-containing products habitually (unless have quit > 4 months prior)
* Current use of medications (except for birth control) or dietary supplements that could alter cardiovascular, thermoregulatory, or vascular control (e.g., anti-hypertensives, statins)
* History of disease of the gastrointestinal tract including (but not limited to) diverticulosis, diverticulitis and inflammatory bowel disease, peptic ulcer disease, Crohn's disease, ulcerative colitis; or previous gastrointestinal surgery
* Have a history of renal disease including (but not limited to) chronic kidney disease, acute kidney injury, kidney stone disease, glomerular disease, or nephritis
* Known allergies to medical adhesives
* Known allergy to MitoQ
* Difficulty swallowing pills
* Heart, lung, kidney, muscle, or nerve disorder(s)
* A planned MRI during the study or within 3 days after completing a cold test
* Women who are pregnant, planning to become pregnant, or breastfeeding
* Not willing to have small areas of skin on the body shaved (if deemed necessary for attachment of study instrumentation)
* Have donated blood within 8 weeks of the study or plan to donate blood during the study
* Lesions on a significant portion of the upper extremities due to skin pigmentation disorders (e.g., vitiligo, psoriasis)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Skin blood flow | Up to 2.5 hours after supplement dose on each cold air exposure and cold water hand immersion study day
  Skin blood flow is measured on the arm, hand, and finger using non-invasive laser probes. Output (red blood cell flux) will be divided by mean arterial blood pressure to give an index of cutaneous vascular conductance [CVC, flux/mmHg].
Body skin temperature | Within 1 hour before and up to 2.5 hours after supplement dose on each cold air exposure and cold water hand immersion study day
  Skin temperatures (°C) at 12 sites on the body will be measured using temperature sensors.

SECONDARY OUTCOMES:
Manual dexterity | Within 1 hour before and approximately 2 hours after supplement dose on each cold air exposure study day
  Manual dexterity is assessed by placing pegs into a pegboard, moving small blocks on a table, and placing bullets into magazines. Scores are the number of pegs placed into the board in 1 minute, the time (seconds) required to move small blocks various distances on the table, and the number of bullets placed into magazines in 2 minutes.
Finger strength | Within 1 hour before and approximately 2 hours after supplement dose on each cold air exposure study day
  Finger strength (kilograms) is measured using a pinch meter. Participants will complete three pinch strength tests on each hand.
Hand strength | Within 1 hour before and approximately 2 hours after supplement dose on each cold air exposure study day
  Hand strength (kilograms) is measured on each hand using a grip strength meter.
Body core temperature | Up to 2.5 hours after supplement dose on each cold air exposure and cold water hand immersion study day
  Body core temperature (°C) is measured using a telemetry pill self-inserted as a suppository or ingested orally.
Metabolic heat production | Up to 2.5 hours after supplement dose on each cold air exposure study day
  Oxygen consumption (liters/minute) and carbon dioxide production (liters/minute) are measured by breathing into a mouthpiece connected to a metabolic cart for ~5 minutes. Oxygen consumption and carbon dioxide production will be combined to report metabolic heat production in Watts per meter squared.
Blood pressure | Up to 2.5 hours after supplement dose on each cold air exposure and cold water hand immersion study day
  Brachial artery blood pressure (mmHg) is measured using an automated cuff.
Heart rate | Up to 2.5 hours after supplement dose on each cold air exposure and cold water hand immersion study day
  Heart rate (beats per minute) is measured using an automated cuff.
Plasma MitoQ | Within 30 minutes before, 1 hour after, and 2.5 hours after supplement dose on each cold air exposure and cold water hand immersion study day
  Circulating concentrations of MitoQ (pmol/milliliter) is assessed in blood collected by venipuncture.
Plasma malondialdehyde | Within 30 minutes before, 1 hour after, and 2.5 hours after supplement dose on each cold air exposure and cold water hand immersion study day
  Circulating concentrations of malondialdehyde (umol/liter) is assessed in blood collected by venipuncture.
Plasma total antioxidant status | Within 30 minutes before, 1 hour after, and 2.5 hours after supplement dose on each cold air exposure and cold water hand immersion study day
  Total antioxidant status (mmol/liter) is assessed in blood collected by venipuncture.
Thermal comfort | Up to 2.5 hours after supplement dose on each cold air exposure and cold water hand immersion study day
  Thermal comfort is assessed using a 1-7 scale (higher number is more discomfort).
Thermal sensation | Up to 2.5 hours after supplement dose on each cold air exposure and cold water hand immersion study day
  Ratings of thermal sensation is assessed using a -50 to 50 scale (50 is extremely hot and -50 is extremely cold).
Pain perception | Up to 2.5 hours after supplement dose on each cold air exposure and cold water hand immersion study day
  Pain is assessed using a 0-10 scale (higher number is more pain).

CONTACTS AND LOCATIONS:
Locations (1):
- U.S. Army Research Institute of Environmental Medicine, Natick, Massachusetts, United States

DOCUMENTS (1):
  • Informed Consent Form (2025-07-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT06784531/ICF_000.pdf